CLINICAL TRIAL: NCT00097110
Title: RCT of Antioxidant Therapy to Prevent Preeclampsia in Brazil
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Global Network for Women's and Children's Health Research (Other); Bill and Melinda Gates Foundation (Other); Fogarty International Center of the National Institute of Health (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Cancer Institute (NCI) (NIH); RTI International (Other); University of Cincinnati (Other); Universidade Federal de Pernambuco (Other); Feculdade de Medicina da Universidade de Sao Paulo - Brasil (Other); Faculdade de Medicina de Botucatu, UNESP, Botucatu, Brasil (Other); University of Campinas, Brazil (Other); Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GN 05; U01HD040565 (NIH)
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Preeclampsia; Eclampsia; HELLP Syndrome; Pregnancy
Keywords: Vitamin C; Vitamin E; Preeclampsia; Antioxidants; Global Network; Preterm birth; Low birth weight infants; Brazil; Brasil; Maternal and child health; International; Women's health
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia; HELLP Syndrome; Premature Birth | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Vitamin C and E

SUMMARY:
The perinatal morbidity and mortality rates for Brazil are five to ten-fold higher than those reported for upper income countries. This study tests the likelihood that the joint administration of antioxidants vitamin C (1000 mg) and vitamin E (400 IU) will reduce the incidence of preeclampsia among chronically hypertensive pregnant patients and patients with a past history of preeclampsia/eclampsia.

DETAILED DESCRIPTION:
The maternal, perinatal and neonatal morbidity and mortality rates for Brazil are five to ten-fold higher than those reported for upper income countries. In Sao Paulo, 22 percent of maternal deaths are attributable to hypertensive complications of pregnancy, which ranks as the number one cause of maternal death. Recent advances in the understanding of the pathophysiology of preeclampsia suggest the possibility of antioxidant therapy for the prevention of preeclampsia. The primary hypothesis is that the joint administration of the antioxidants vitamin C (1000 mg) and vitamin E (400 IU) will reduce the incidence of preeclampsia among chronically hypertensive pregnant patients and patients with a past history of preeclampsia/eclampsia. Secondary outcomes include severity of preeclampsia; incidence of gestational hypertension; incidence of premature rupture of the membranes; incidence of preterm birth; incidence of low birth weight infants; biomarker level correlation with preeclampsia.

Study sites are high-risk obstetrical clinics in the Brazilian cities of Recife, Botucatu, Campinas, and Porto Alegre. The sample size was based on an estimated risk of preeclampsia/eclampsia of 21-25% in the control group. The study hypothesizes a 40% absolute reduction of risk of preeclampsia; early treatment withdrawal of 3%; withdrawal of consent or loss to follow-up of 10%; calculated at a 0.05 significance level with 80% power. Seven hundred thirty-four obstetric patients with chronic hypertension or preeclampsia in the prior pregnancy presenting for care between 12 weeks and 19 weeks', 6 days gestation will be randomized to a double-blinded placebo controlled trial to receive a daily dose of either vitamin E (400 International Units) and vitamin C (1000 mg) or placebo from the time of enrollment to delivery. The use of MEMS caps enables researchers to accurately track compliance.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 12 weeks and 19 weeks, 6 days, inclusive
* Chronic hypertension
* History of preeclampsia/eclampsia
* Attendance at a participating hospital (Recife, Botucatu, Campinas and Porto Alegre, Brazil)

Exclusion Criteria:

* Planned delivery elsewhere.
* Multifetal gestation.
* Allergy to vitamin C or vitamin E.
* Requirement for aspirin or anticoagulant medication.
* Proteinuria ≥ 2+ on dipstick urine test; or proteinuria = 1+ on dipstick and ≥ 300 mg/24 hours.
* Pre-pregnancy diabetes mellitus.
* Known fetal anomaly incompatible with life.
* Prior participation in the study.
* Unwillingness to take the study medication.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 734
Dates: Start 2003-07; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Incidence of preeclampsia

SECONDARY OUTCOMES:
Severity of preeclampsia
Incidence of gestational hypertension or preeclampsia
Frequency of abruptio placentae
Incidence of preterm birth
Incidence of small for gestational age
Incidence of low birth weight infants
Biomarker level correlation with preeclampsia

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A. Spinnato, M.D., Principal Investigator — University of Cincinnati
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Spinnato JA 2nd, Freire S, Pinto e Silva JL, Rudge MV, Martins-Costa S, Koch MA, Goco N, Santos Cde B, Cecatti JG, Costa R, Ramos JG, Moss N, Sibai BM. Antioxidant supplementation and premature rupture of the membranes: a planned secondary analysis. Am J Obstet Gynecol. 2008 Oct;199(4):433.e1-8. doi: 10.1016/j.ajog.2008.07.011. PMID 18928997
- [Derived] Spinnato JA 2nd, Freire S, Pinto E Silva JL, Cunha Rudge MV, Martins-Costa S, Koch MA, Goco N, Santos Cde B, Cecatti JG, Costa R, Ramos JG, Moss N, Sibai BM. Antioxidant therapy to prevent preeclampsia: a randomized controlled trial. Obstet Gynecol. 2007 Dec;110(6):1311-8. doi: 10.1097/01.AOG.0000289576.43441.1f. PMID 18055726
- See also: Global Network for Women's and Children's Health Research — http://gn.rti.org
- See also: RTI International — http://www.rti.org/